CLINICAL TRIAL: NCT03616834
Title: Tomivosertib (eFT-508) in Combination With PD-1/PD-L1 Inhibitor Therapy: A Study of Subjects Administered Anti-PD-1/Anti-PD-L1 Therapy That Are Experiencing Insufficient Response to Checkpoint Inhibitor Alone
Brief Title: Tomivosertib (eFT-508) in Combination With PD-1/PD-L1 Inhibitor Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Effector Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eFT508-0010
Record Dates: First submitted 2018-07-09; First posted 2018-08-06 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2019-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — tomivosertib

STUDY DESIGN:
Intervention Model Description: Subjects will continue their anti-PD-1/anti-PD-L1 therapy, which they had already initiated per standard of care according to the package insert, and then initiate Tomivosertib (eFT-508) at 200 mg twice daily (bid) 7 days prior to their next scheduled anti-PD-1/anti-PD-L1 therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tomivosertib (eFT-508) (Experimental): Tomivosertib (eFT-508) will be taken at 200 mg twice daily (bid). Subjects will continue their anti-PD-1/anti-PD-L1 therapy, which they had already initiated per standard of care according to the package insert.
  Interventions: Drug: Tomivosertib (eFT-508)

INTERVENTIONS:
Drug: Tomivosertib (eFT-508) — Tomivosertib (eFT-508) is a novel, small-molecule investigational drug being developed by eFFECTOR Therapeutics, as an antitumor therapy that acts by selectively inhibiting mitogen-activated protein kinase (MAPK)-interacting serine/threonine kinase (MNK)1 and MNK 2.
  Other Names: MNK1 and MNK2

SUMMARY:
Phase 2, open-label study that will evaluate the safety, tolerability, antitumor activities.

DETAILED DESCRIPTION:
This Phase 2, open-label study will evaluate the safety, tolerability, antitumor activity, and pharmacokinetics (PK) of Tomivosertib (eFT-508) in subjects who have initiated anti-PD-1/anti-PD-L1 monotherapy and either developed progressive disease (PD) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 on therapy or have undergone 12 weeks of anti-PD-1/anti-PD-L1 therapy with no evidence of partial response (PR) or complete response (CR).

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent and any authorizations required by local law;
* Men or women 18 years of age;
* Initiated monotherapy with an anti-PD-1 or anti-PD-L1 agent (avelumab, atezolizumab, durvalumab, nivolumab, or pembrolizumab) in accordance with the package insert, and:
* Are judged by the Principal Investigator as tolerating the anti-PD-1 or anti-PD-L1 therapy, and
* Developed PD per RECIST 1.1 on therapy, or
* Have undergone 12 weeks of anti-PD-1 or anti-PD-L1 therapy with no evidence of PR or CR;
* ECOG performance status of 0 or 1;
* Has at least 1 measurable lesion per RECIST 1.1 criteria;
* Adequate bone marrow function during Screening as defined below:
* Absolute neutrophil count 1.0 109/L,
* Platelet count 75 109/L, and
* Hemoglobin 80 g/L (8.0 g/dL or 4.9 mmol/L);
* Adequate hepatic function during Screening as defined below:
* Serum alanine aminotransferase 3 upper limit of normal (ULN) or 5 ULN if liver metastases are present,
* Serum aspartate aminotransferase 3 ULN or 5 ULN if liver metastases are present, and
* Serum bilirubin - total 1.5 ULN (unless due to Gilbert's syndrome or hemolysis);
* Adequate renal function during Screening, defined as measured or estimated creatinine clearance 60 mL/min calculated by the Cockcroft-Gault formula using actual body weight;
* Adequate coagulation profile during Screening as defined below:
* Prothrombin time within the ULN, and
* Activated partial thromboplastin time within the ULN;
* Negative antiviral serology during Screening as defined below:
* Negative human immunodeficiency virus antibody,
* Negative hepatitis B surface antigen and negative hepatitis B core antibody or undetectable hepatitis B virus (HBV) DNA by quantitative polymerase chain reaction (qPCR) testing. Note: Hepatocellular carcinoma (HCC) subjects with - -- HBV may only be enrolled if their hepatitis is judged clinically stable by the Investigator, and
* Negative hepatitis C virus (HCV) antibody or negative HCV ribonucleic acid by q PCR. Note: HCC subjects with HCV are permitted provided they are not being actively treated;
* Female subjects of childbearing potential must meet all of the following criteria:
* Not pregnant (negative serum pregnancy test during Screening),
* Not breastfeeding, and
* Willing to use a protocol-recommended method of contraception or to abstain from heterosexual intercourse from the start of Tomivosertib (eFT-508) until at least 30 days after the last dose of Tomivosertib (eFT-508) or anti-PD-1/anti-PD-L1 therapy. Note: A female subject is considered to be of childbearing potential unless she has had a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy; has medically documented ovarian failure (with serum estradiol and follicle-stimulating hormone levels within the institutional laboratory postmenopausal range and a negative serum or urine beta human chorionic gonadotropin); or is menopausal (age 55 years with amenorrhea for 6 months);
* Male subjects who can father a child must meet all of the following criteria:
* Willing to use a protocol-recommended method of contraception or to abstain from heterosexual intercourse with females of childbearing potential from the start of Tomivosertib (eFT-508) until at least 30 days after the last dose of Tomivosertib (eFT-508) or anti-PD-1/anti-PD-L1 therapy, and
* Willing to refrain from sperm donation from the start of Tomivosertib (eFT-508) until at least 90 days after the last dose of Tomivosertib (eFT-508) or anti-PD-1/anti-PD-L1 therapy. Note: A - male subject is considered able to father a child unless he has had a bilateral vasectomy with documented aspermia or a bilateral orchiectomy;
* Willing to comply with the scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions. Note: Psychological, social, familial, or geographical factors that might preclude adequate study participation should be considered;
* In the judgment of the Investigator, participation in the protocol offers an acceptable benefit-to-risk ratio when considering current disease status, medical condition, and the potential benefits and risks of alternative treatments for the subject's cancer; and
* Estimated life expectancy of 3 months.

Exclusion Criteria:

* Currently in CR or PR with anti-PD-1 or anti-PD-L1 monotherapy (avelumab, atezolizumab, durvalumab, nivolumab, or pembrolizumab);
* History of another malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin; in situ cervical carcinoma; adequately treated, papillary, noninvasive bladder cancer; other adequately treated Stage 1 or 2 cancers currently in complete remission; or any other cancer that has been in complete remission for 2 years
* Gastrointestinal (GI) disease (eg, gastric or intestinal bypass surgery, pancreatic enzyme insufficiency, malabsorption syndrome, symptomatic inflammatory bowel disease, chronic diarrheal illness, bowel obstruction) that may interfere with drug absorption or with interpretation of GI AEs;
* Known symptomatic brain metastases requiring 10 mg/day of prednisolone (or its equivalent). Subjects with previously diagnosed brain metastases are eligible if they have completed their treatment, have recovered from the acute effects of radiation therapy or surgery prior to the start of Tomivosertib (eFT-508), fulfill the steroid requirement for these metastases, and are neurologically stable;
* Significant cardiovascular disease, including myocardial infarction, arterial thromboembolism, or cerebrovascular thromboembolism, within 6 months prior to start of Tomivosertib (eFT-508); symptomatic dysrhythmias or unstable dysrhythmias requiring medical therapy; angina requiring therapy; symptomatic peripheral vascular disease; New York Heart Association Class 3 or 4 congestive heart failure; Grade 3 hypertension (diastolic blood pressure 100 mmHg or systolic blood pressure 160 mmHg); or history of congenital prolonged QT syndrome;
* Significant ECG abnormalities at Screening, including unstable cardiac arrhythmia requiring medication, left bundle branch block, second-degree atrioventricular (AV) block type II, third-degree AV block, Grade 2 bradycardia, or QT interval corrected using Fridericia's formula >450 msec (for men) or >470 msec (for women);
* Ongoing risk for bleeding due to active peptic ulcer disease or bleeding diathesis;
* Evidence of an ongoing systemic bacterial, fungal, or viral infection (including upper respiratory tract infections) at the start of Tomivosertib (eFT-508). Note: Subjects with localized fungal infections of skin or nails are eligible. Subjects may be receiving prophylactic antibiotics as long as the antibiotic is not prohibited by the protocol due to the potential for drug-drug interactions;
* Has received a live vaccine within 30 days of planned start of Tomivosertib (eFT-508);
* Pregnant or breastfeeding;
* Major surgery within 4 weeks before the start of Tomivosertib (eFT-508);
* Prior solid organ or bone marrow progenitor cell transplantation;
* Prior therapy with any known inhibitor of MNK1 or MNK2;
* Prior high-dose chemotherapy requiring stem cell rescue;
* History of or active autoimmune disorders or other conditions that might impair or compromise the immune system;
* Any prior exposure to cytotoxic T-lymphocyte-associated protein 4 inhibitors;
* Ongoing immunosuppressive therapy, including systemic or enteric corticosteroids. Note: At Screening and during study participation, subjects may be using systemic corticosteroids (doses 10 mg of prednisone or equivalent) or topical or inhaled corticosteroids;
* Use of a strong inhibitor or inducer of cytochrome P450 (CYP)3A4 within 7 days prior to the start of Tomivosertib (eFT-508) or expected requirement for use of a strong CYP3A4 inhibitor or inducer during study participation; Need for proton pump inhibitors and histamine H2 blockers at study entry;
* Previously received investigational product in a clinical trial within 30 days or within 5 elimination half-lives (whichever is longer) prior to the start of Tomivosertib (eFT-508), or is planning to take part in another clinical trial while participating in this study;
* Has any illness, medical condition, organ system dysfunction, or social situation, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a subject's ability to sign Informed - Consent Document(s), adversely affect the subject's ability to cooperate and participate in the study, or compromise the interpretation of study results;
* Portal vein invasion at the main portal (Vp4), inferior vena cava, or cardiac - involvement of HCC based on imaging; or
* Has had esophageal or gastric variceal bleeding within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with treatment-emergent AEs (TEAEs) and serious AEs (SAEs) | 52 weeks
  The incidence of TEAEs and SAEs will be summarized and TEAEs will also be summarized by severity and according to their relationship to Tomivosertib (eFT-508).
Overall Response Rate (ORR) as determined by RECIST 1.1 | 52 weeks
  Defined as the proportion of subjects who achieve a best overall response of complete response (CR) or partial response (PR).
Progression Free Survival (PFS) as determined by RECIST 1.1 | 52 weeks
  Defined as the interval from the start of Tomivosertib (eFT-508) to the occurrence of PD or death from any cause.

SECONDARY OUTCOMES:
ORR as determined by iRECIST | 52 weeks
  Defined as the proportion of subjects who achieve a best overall response of CR assigned using iRECIST (iCR) or PR assigned using iRECIST (iPR).
PFS as determined by iRECIST | 52 weeks
  Defined as the interval from the start of Tomivosertib (eFT-508) to the occurrence of confirmed progression assigned using iRECIST (iCPD) or death from any cause.
Overall survival | 52 weeks
  Defined as time from the first dose date of Tomivosertib (eFT-508) to death due to any cause will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Lyon Gleich, MD, Study Director — Medpace, Inc.
Locations (19):
- United States (19):
  - University of Arizona - Cancer Center, Tucson, Arizona
  - Pacific Shores Medical Group, Long Beach, California
  - Hoag Memorial Hospital Presbyterian, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - St. Mary's Medical Center, San Francisco, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Columbus Regional Research Institute, Columbus, Georgia
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Indiana University Health Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Gabrail Cancer Center, Canton, Ohio
  - Universty of Toledo Medical Center, Toledo, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Oncology Consultants, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lucibello G, Mograbi B, Milano G, Hofman P, Brest P. PD-L1 regulation revisited: impact on immunotherapeutic strategies. Trends Mol Med. 2021 Sep;27(9):868-881. doi: 10.1016/j.molmed.2021.06.005. Epub 2021 Jun 26. PMID 34187739